CLINICAL TRIAL: NCT03659279
Title: Pilot Study of "Let's Get Organized" - a Group Intervention for Improving Time Management
Brief Title: Let's Get Organized Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: Dalarna County Council, Sweden (Other); Region Örebro County (Other); Uppsala University (Other); Region Gävleborg (Other); State University of New York - Downstate Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORU 2015/015
Record Dates: First submitted 2018-08-20; First posted 2018-09-06 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Neurodevelopmental Disorders; Mental Disorder
Keywords: Time management; Group intervention; Executive function
MeSH Terms: conditions — Neurodevelopmental Disorders; Mental Disorders

STUDY DESIGN:
Intervention Model Description: Pre-post intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Let's Get Organized (Experimental): Group intervention with 10 weekly sessions, each lasting 1.5 hours.
  Interventions: Behavioral: Let's Get Organized

INTERVENTIONS:
Behavioral: Let's Get Organized — Group intervention aiming to enhance time-management, targeted to persons with mental or neurodevelopment disorders. Each group has 6-8 participants and is lead by two trained group leaders. Goal-directed and other learning strategies are used to train effective time management habits such as maintaining a calendar and wearing a watch. Group sessions are structured with a PowerPoint presentation and a course manual, and information from the group leaders is intermixed with discussion among the participants and tasks to complete.
  Other Names: LGO

SUMMARY:
The aim of this study is to pilot test the Let's Get Organized (LGO) Occupational Therapy intervention in a Swedish context by exploring possible enhancements in time management skills, aspects of executive functioning, and satisfaction with daily occupations in persons with time-management difficulties due to neurodevelopmental and/or mental disorders.

Method:

A pre-post design with 3 and 12-months follow-up is used.

The LGO intervention is a manual-based group intervention aiming to enhance time-management, targeted to persons with mental or neurodevelopmental disorders. The LGO is conducted as 10 weekly 1.5-hour group sessions. Two trained group leaders, lead each group of 6-8 participants. Goal-directed and other learning strategies are used to train effective time management habits such as maintaining a calendar and wearing a watch. All group sessions follow the same format, and each session has a set theme. Group sessions are structured with a slide presentation and a course manual, and information from the group leaders is intermixed with discussion among the participants and tasks to complete.

The primary outcome of the study is self-reported time management measured by the Assessment of Time Management Skills (ATMS-S). Secondary outcomes are executive functioning measured with the Weekly Calendar Planning Activity (WCPA) and satisfaction with daily occupations, which is measured with the interview-administered questionnaire Satisfaction with Daily Occupations 13 items (SDO-13).

Data will be collected before intervention start (pre intervention), after intervention completion (post intervention) and 3 and 12 months post intervention completion. The ATMS will be collected at all four time points. The WCPA and SDO-13 will be collected pre, post and 12 months post intervention.

ELIGIBILITY:
Inclusion Criteria:

* confirmed or suspected diagnosis of a mental disorder, such as affective disorder or schizophrenia, or neurodevelopmental disorder, such as autism spectrum disorder or attention deficit hyperactivity disorder/attention deficit disorder
* self-reported difficulties in time management in daily life to an extent that affects functioning in daily life negatively

Exclusion Criteria:

* intellectual disability

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change Assessment of Time Management Skills (ATMS-S) Time management sub scale | baseline (pre-intervention), 10 weeks, 24 weeks, 62-months
  Time management (11 items) measured in ATMS units (range 0-100)

SECONDARY OUTCOMES:
Change in Weekly Calendar Planning Activity (WCPA-SE) No of appointments | baseline (pre-intervention), 10 weeks, 62-months
  No of correctly entered appointments (range 0-17) Total time No of strategies used No of rules followed (0-5)
Change in Weekly Calendar Planning Activity (WCPA-SE) Total time | baseline (pre-intervention), 10 weeks, 62-months
  Total time No of strategies used No of rules followed (0-5)
Change in Weekly Calendar Planning Activity (WCPA-SE) Strategies | baseline (pre-intervention), 10 weeks, 62-months
  No of strategies used No of rules followed (0-5)
Change in Weekly Calendar Planning Activity (WCPA-SE) Rules followed | baseline (pre-intervention), 10 weeks, 62-months
  No of rules followed (range 0-5)
Change in Satisfaction with Daily Occupations 13 items (SDO-13) Activity sub scale | baseline (pre-intervention), 10 weeks, 62-months
  No of activities (range 0-13)
Change in Satisfaction with Daily Occupations 13 items (SDO-13) Satisfaction sub scale | baseline (pre-intervention), 10 weeks, 62-months
  Satisfaction sub scale score (each item is scored 1-7 and summed to a sub scale score, range 13-91, higher score indicates better satisfaction)
Change in Satisfaction with Daily Occupations 13 items (SDO-13) Global satisfaction sub scale | baseline (pre-intervention), 10 weeks, 62-months
  Global satisfaction score (range 1-5, lower score indicates better satisfaction)
Change in Assessment of Time Management Skills (ATMS-S) Organization and planning sub scale | baseline (pre-intervention), 10 weeks, 24 weeks, 62-months
  Organization and Planning (11 items) measured in ATMS units (range 0-100)
Change in Assessment of Time Management Skills (ATMS-S) Regulation of emotions sub scale | baseline (pre-intervention), 10 weeks, 24 weeks, 62-months
  Regulation of emotions (5 items) measured in ATMS units (range 0-100)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Holmefur, PhD, Principal Investigator — Örebro University, Sweden

IPD SHARING:
Plan to Share IPD: No